CLINICAL TRIAL: NCT00486252
Title: Non Interventional Study in Patients With Open Angle Glaucoma and/or Ocular Hypertension Treated With XALATAN® (Latanoprost) as First-Line Monotherapy and as Second-Line Monotherapy After Beta-Blockers Therapy Failure
Brief Title: Non Interventional Study in Patients With Open Angle Glaucoma and/or Ocular Hypertension Treated With XALATAN®
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A6111138
Record Dates: First submitted 2007-06-12; First posted 2007-06-14 (Estimated); Results first posted 2009-07-16 (Estimated); Last update posted 2021-03-01 (Actual); Status verified 2009-11

CONDITIONS: Glaucoma,Open-Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- This is N/A due to the above description.: This is N/A due to the above description.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — This is a non-interventional study. Subgroups of naïve patients and patients with previous failure to beta-blockers therapy were analyzed.

SUMMARY:
The primary objective is to evaluate the Intraocular pressure reducing effect of Xalatan over 3 months. The secondary objective is to study the other efficacy parameters during treatment for 3 months

ELIGIBILITY:
Inclusion Criteria:

* Unilateral or bilateral open angle glaucoma or ocular hypertension (IOP (Intraocular Pressure) ≥ 21 mmHg at diagnosis).
* Naive patients (no prior anti-glaucoma pharmacological or surgical treatment) and patients with beta-blockers therapy failure
* Visual acuity (best corrected) equal to or better than 6/6

Exclusion Criteria:

* closed/barely open anterior chamber angle or history of acute angle closure glaucoma.
* history of any antiglaucoma surgical treatment (Argon Laser Trabeculoplasty and/or any ocular filtering surgical intervention).
* ocular surgery (on the globe of the eye only), or inflammation/infection within 3 months prior to baseline visit. (Applies to both fellow and study eyes.)
* other abnormal ocular conditions or symptoms preventing the patient from entering the study, in the investigator's clinical judgement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: outpatients with unilateral or bilateral open angle glaucoma or ocular hypertension
Sampling Method: Non-Probability Sample
Enrollment: 996 (Actual)
Dates: Start 2007-06; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6111138&StudyName=Non%20Interventional%20Study%20in%20Patients%20with%20Open%20Angle%20Glaucoma%20and/or%20Ocular%20Hypertension%20Treated%20with%20XALATAN%AE%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Latanoprost All Subjects: Subjects administered 1 drop of latanoprost (0.005%, 50 μg/mL) eye drops solution daily as prescribed by the investigator.
Period: Overall Study
Arm/Group | Latanoprost All Subjects
Started | 996
Completed | 938
Not Completed | 58
Not completed — Adverse Event | 7
Not completed — Lack of Efficacy | 9
Not completed — Lost to Follow-up | 24
Not completed — Other | 18

BASELINE CHARACTERISTICS:
Arm/Group | Latanoprost All Subjects
Number analyzed (Participants) | 996
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (13.4)
Sex/Gender, Customized [Number; unit: participants]
  Male | 395
  Female | 596
  Unspecified | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Intraocular Pressure (IOP): Baseline to Month 3
Description: Change: IOP at observation minus IOP at baseline. IOP was measured with the non-contact or Goldmann tonometer for a given subject. Three measurements were performed in each eye alternating between the eyes, starting with the right eye. The mean of the 3 measurements was used and if both eyes were study eyes, the mean of the 2 eyes was used.
Time Frame: Baseline, Month 3
Population: Full Analysis Set (FAS) included all patients who received at least 1 dose of latanoprost (Xalatan®), had baseline IOP recorded, & at least one postbaseline IOP measure recorded (at either Month 1 or Month 3). No imputation techniques used for missing data; only observed data reported. "n"=number of participants in each group for that category.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Latanoprost (All Subjects): Subjects administered 1 drop of latanoprost (0.005%, 50 μg/mL) eye drops solution daily as prescribed by the investigator.
- Latanoprost (no Prior Beta-blocker Therapy): Naive Subject: Subjects with no prior beta-blocker therapy were administered 1 drop of latanoprost (0.005%, 50 μg/mL) eye drops solution daily as prescribed by the investigator.
- Latanaprost (Prior Beta-blocker Failure): Subjects previously receiving beta-blocker: Subjects who previously failed beta-blocker therapy were administered 1 drop of latanoprost (0.005%, 50 μg/mL) eye drops solution daily as prescribed by the investigator.
Arm/Group | Latanoprost (All Subjects) | Latanoprost (no Prior Beta-blocker Therapy) | Latanaprost (Prior Beta-blocker Failure)
Number analyzed (Participants) | 945 | 402 | 531
mmHg | -5.3 (3.9) | -6.8 (3.8) | -4.1 (3.5)

2. Secondary Outcome: Percentage Change in Intraocular Pressure (IOP)
Description: Percentage change in IOP calculated as 100 times (IOP at Observation minus IOP at Baseline) divided by IOP at Baseline.
Time Frame: Month 1, Month 3
Population: Full Analysis Set (FAS) included all patients who received at least 1 dose of latanoprost (Xalatan®), had baseline IOP recorded, & at least one postbaseline IOP measure recorded (at either Month 1 or Month 3). No imputation techniques used for missing data; only observed data reported.
Measure: Mean (Standard Deviation); unit: percentage change in mmHg
Arm/Group | Latanoprost (All Subjects) | Latanoprost (no Prior Beta-blocker Therapy) | Latanaprost (Prior Beta-blocker Failure)
Number analyzed (Participants) | 945 | 402 | 531
percentage change in mmHg
  Month 1 (n=982, 419, 551) | -19.2 (20.9) | -22.6 (28.0) | -16.5 (12.7)
  Month 3 (n=945, 402, 531) | -21.5 (22.2) | -26.1 (29.0) | -18.1 (14.5)

3. Secondary Outcome: Categorized Percentage Change in Intraocular Pressure (IOP)
Description: Percentage change=100 times (IOP at observation minus IOP at Baseline) divided by IOP at Baseline. Percentage change in each patient assigned to the following: Increase or no change in IOP (percentage change greater than or equal to 0); Percentage reduction of up to 20% (-20 less than or equal to percentage change < 0); Percentage reduction greater than 20% (percentage change < -20).
Time Frame: Month 1, Month 3
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Latanoprost (All Subjects) | Latanoprost (no Prior Beta-blocker Therapy) | Latanaprost (Prior Beta-blocker Failure)
Number analyzed (Participants) | 990 | 422 | 556
participants
  Month 1: Increase or no change in IOP | 69 | 10 | 58
  Month 1: Percentage reduction of up to 20% | 422 | 145 | 274
  Month 1: Percentage reduction of greater than 20% | 491 | 264 | 219
  Month 3: Increase or no change in IOP | 62 | 12 | 50
  Month 3: Percentage reduction of up to 20% | 312 | 90 | 217
  Month 3: Percentage reduction of greater than 20% | 571 | 300 | 264

4. Other Pre Specified Outcome: Change in Intraocular Presssure (IOP): Baseline to Month 1
Description: Change: IOP at observation minus IOP at baseline. IOP was measured with the non-contact or Goldmann tonometer for a given subject. Three measurements were performed in each eye alternating between eyes, starting with the right eye. The mean of the 3 measurements was used and if both eyes were study eyes, the mean of the 2 eyes was used.
Time Frame: Baseline, Month 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Latanoprost (All Subjects) | Latanoprost (no Prior Beta-blocker Therapy) | Latanaprost (Prior Beta-blocker Failure)
Number analyzed (Participants) | 982 | 419 | 551
mmHg | -4.7 (3.4) | -5.9 (3.5) | -3.7 (3.0)

ADVERSE EVENTS:
Arm/Group | Latanoprost All Subjects
Serious Adverse Events (participants affected / at risk) | 0/996
Other Adverse Events (participants affected / at risk) | 122
OTHER ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Latanoprost All Subjects
Abnormal sensation in eye (Eye disorders) | 1/996
Conjunctival hyperaemia (Eye disorders) | 11/996
Conjunctival irritation (Eye disorders) | 1/996
Conjunctival oedema (Eye disorders) | 1/996
Conjunctival pigmentation (Eye disorders) | 1/996
Conjunctivitis (Eye disorders) | 3/996
Dry eye (Eye disorders) | 1/996
Erythema of eyelid (Eye disorders) | 4/996
Eye irritation (Eye disorders) | 1/996
Eye pain (Eye disorders) | 1/996
Eyelash discolouration (Eye disorders) | 2/996
Keratoconjunctivitis sicca (Eye disorders) | 1/996
Sicca syndrome (Eye disorders) | 2/996
Visual disturbance (Eye disorders) | 1/996
Adverse event (General disorders) | 34/996
Blood pressure decreased (Investigations) | 1/996
Headache (Nervous system disorders) | 1/996
Paraesthesia (Nervous system disorders) | 1/996
Hyperaemia (Vascular disorders) | 62/996

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of <60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), <12 mo from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.